# TRANSCENDENCE RESEARCH: Holistic Education For Colonized Countries Primarily English Speaking

NCT06098755

January 24, 2026



# **Understanding SOAP Notes**

SOAP notes are a standardized method of documentation used to record and communicate patient information. This structured format ensures that essential details are captured in a clear, concise, and organized manner, facilitating continuity of care and informed decision-making.

# **SOAP Breakdown**

## S - Subjective

- Represents the *client*'s perspective.
- Includes their feelings, concerns, and goals.
- Direct quotes can be valuable.
- Examples:
  - o "I've been feeling anxious all week."
  - "Our sessions are really helping me."

#### A - Assessment

- The *therapist*'s professional analysis of the subjective and objective information.
- Includes progress, insights, and any changes in the client's condition.
- Examples:
  - Client is showing progress in managing anxiety symptoms.
  - Potential for increased self-awareness observed.

## O - Objective

- Represents the therapist's observations.
- Includes factual information, such as behavior and appearance.
- Avoid personal opinions or interpretations.
- Examples:
  - Client appeared agitated during the session.
  - Client maintained good eye contact.

## P - Plan

- Outlines the therapist's future actions and interventions.
- Includes goals for the next session and adjustments to treatment.
- Examples:
  - Continue to explore coping mechanisms for anxiety.
  - Introduce mindfulness exercises.

#### SOAP notes are critical for:

- Continuity of Care: Ensuring that all therapists involved have a clear understanding of the client's history and progress.
- Legal Protection: Providing a detailed record of treatment in case of legal or ethical inquiries.

- **Treatment Planning:** Informing the therapist's decisions about future sessions and interventions.
- **Communication:** Facilitating communication among healthcare providers, when necessary and with appropriate consent.
- Quality Assurance: Supporting the evaluation and improvement of therapy services.

By consistently using the SOAP note format, psychotherapists can enhance the quality and effectiveness of their documentation, ultimately benefiting both themselves and their clients.

- SOAP notes offer a structured way to document therapy sessions.
- Each section (Subjective, Objective, Assessment, Plan) captures different but vital information.
- They promote clear communication, legal protection, and effective treatment planning.
- Regular use improves the quality of care and therapeutic outcomes.